CLINICAL TRIAL: NCT00910949
Title: Chronic Pain After Thoracotomy
Brief Title: Sensory Perception After Thoracotomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: MD, Kim Wildgaard, Section for Surgical Pathophysiology 4074
Other Study IDs: H-B-2008-059b
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Neuropathic Pain; Thoracotomy; Chronic Pain
Keywords: persistent pain; neuropathic pain; Thoracotomy; Chronic Pain
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Painfree: Thoracotomy patients without chronic pain
- With Pain: Thoracotomy patients with chronic pain

SUMMARY:
The study will investigate characteristics of chronic pain after thoracotomy

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give consent
* Can read
* Residing in Denmark

Exclusion Criteria:

* Unable to understand the written information in Danish
* Abuse (Medicine, Drugs, Alcohol)
* Severe psychiatric Illness
* Conflicting neurological disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
QST score | 1 y

CONTACTS AND LOCATIONS:
Locations (1):
- Section for Surgical Pathophysiology 4074, Copenhagen, Denmark

REFERENCES:
- [Background] Wildgaard K, Ravn J, Kehlet H. Chronic post-thoracotomy pain: a critical review of pathogenic mechanisms and strategies for prevention. Eur J Cardiothorac Surg. 2009 Jul;36(1):170-80. doi: 10.1016/j.ejcts.2009.02.005. PMID 19307137